CLINICAL TRIAL: NCT05080985
Title: Paravertebral Block Versus Erector Spinae Plane Block for Analgesia and Opioid Consumption in Modified Radical Mastectomy; Randomized, Prospective, Double Blind
Brief Title: Paravertebral Block Versus Erector Spinae Plane Block for Analgesia in Modified Radical Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Nukhet Sivrikoz, Attending Anesthesiologist, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-1608
Record Dates: First submitted 2021-09-15; First posted 2021-10-18 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Postoperative Pain
Keywords: Acute postoperative pain; Nerve block; Thoracic wall
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group P : TPVB (Experimental): Thoracic paravertebral block
  Interventions: Procedure: TPVB; Drug: Bupivacain
- Group E : ESPB (Experimental): Erector spinae plane block
  Interventions: Procedure: ESPB; Drug: Bupivacain

INTERVENTIONS:
Procedure: TPVB — 20 ml 0.375 % bupivacaine was injected between superior costotransverse ligament and pleura.
  Arms: Group P : TPVB
Procedure: ESPB — 20 ml 0.375 % bupivacaine was injected between deep fascia of the erector spinae muscle and transverse process.
  Arms: Group E : ESPB
Drug: Bupivacain — 20 ml 0.375 % bupivacaine was injected

SUMMARY:
The study is planned to be a single-center randomized, prospective double-blind study and includes patients who planned to be done unilateral MRM (modified radical mastectomy) operation in Istanbul University Istanbul Faculty of Medicine. The objective of this study is to compare postoperative analgesic efficacies of TPVB (thoracic paravertebral block) and ESPB (erector spinae plane block) performed under ultrasound (USG) guidance after MRM. Primary outcome of this study is postoperative 24-hour morphine consumption whereas secondary outcomes were planned as the comparison of changes in hemodynamic parameters and numeric rating pain score (NRS).

DETAILED DESCRIPTION:
A total of 86 patients were randomized into TPVB (Group P) and ESPB (Group E) by using closed envelopes.

All patients in the operating room has same anesthetic management under standard monitoring modalities. Prior to regional technique, mild sedation was achieved with midazolam (1-2 mg) and fentanyl (50 mcg). Both blocks were performed under ultrasonography guidance from the level of T4 vertebra with a linear probe (5MHz; GE Healthcare, Wauwatosa, Wis, USA) using longitudinally out-of-plane technique by an anesthesiologist. A 22-gauge, 50 mm insulated stimulating needle was used.By using reference points of C7 and T7, spinous processes of thoracic vertebras were marked. 10% povidone iodine was used for skin antisepsis. USG probe was longitudinally placed at the level of T4. Staff anesthesiologist had to visualize of adjacent muscles, transverse process (TP) and pleura.

For ESPB; confirmation of the needle position was achieved with spread of 2 ml saline between the deep fascia of the erector spinae muscle and the TP. After negative aspiration 20 ml 0.375% bupivacaine was injected with appropriate distribution of LA.

For TPVB; the needle was advanced passing over superior costotransverse ligament and target space was confirmed by the downward displacement of pleura after the administration of 2 ml 0.9% NaCl. After negative aspiration, 20 ml 0.375 % bupivacaine was injected with appropriate distribution of local anesthetics.

Vascular puncture, haematoma, neuraxial injury and pneumothorax were defined as block complications and should be noted.

30 minutes after the block achieved, pinprick test was performed on both mid-axillary and midclavicular lines from T1 to T12 (0 there is sensation, 1 decreased sensation, 2 there is no sensation).

Anesthesia induction was unique for all patients with 0.03 mg kg-1 midazolam, 0.5 mcg kg-1 fentanyl, 2 mg kg-1 propofol and 0.6 mg kg-1 rocuronium. Maintenance was achieved with sevoflurane of 1 minimum alveolar concentration in a mixture of 40% O2 and 60% N2O. As a component of multimodal analgesia, paracetamol (1 gr) was applied to all patients before skin incision.

Hemodynamic data were recorded throughout surgery. An increase more than 20% from baseline in mean arterial pressure (MAP) was defined as inadequate analgesia and was treated with bolus fentanyl (50 mcg). Hypotension was described with a decrease more than 20% in MAP and treated with ephedrine bolus. Bradycardia was determined with a heart rate (HR) less than 50 beats min-1 and treated with atropine. At the end of surgery, the patients were extubated in operating room.

Postoperative analgesia was achieved with IV morphine via Patient Controlled Analgesia (PCA) for 24 hours (0.01 mg kg-1 h-1 basal infusion, 1 mg bolus, 20 minutes lock-out time).

Postoperative follow-up included hemodynamic variables as well as pain scores and morphine consumption. Adequate analgesia at rest (static) and at moving of the arm interpreted as 45-90 degree abduction (dynamic) was investigated with Numeric Rating Scale (NRS) at 30th minute and 1st, 4th, 6th, 12th, 24th hours postoperatively. When NRS was 4 and higher, tramadol should be administered as rescue analgesic. In case of insufficient pain control at 30th minute, dermatomal analgesia should be assessed for both mid-axillary and midclavicular lines from T1 to T8 by pinprick test (0 there is sensation, 1 decreased sensation, 2 there is no sensation). Morphine consumption was evaluated at same study times.

Complications were determined as sedation assessed by Ramsey scale, postoperative nausea- vomiting (PONV) assessed with the four-point categorical scale (0=no PONV, 1=mild nausea, 2=severe nausea or vomiting once, and 3=vomiting more than once). Severe vomiting should be treated in a multimodal way and excluded from the study (category 2,3).

Staff anesthesiologist responsible for operative course did not contribute in analgesia assessment, nor in other postoperative follow-up. Other investigators who were blinded to operative management, collected postoperative data.

ELIGIBILITY:
Inclusion Criteria:

* unilateral MRM
* ages 18-75 years
* American Society of Anesthesiologists (ASA) classification I-III

Exclusion Criteria:

* presence of contraindications for using regional anesthesia (not having patient approval, presence of bleeding-clotting disorders, infection at the injection site, local anesthetic allergy)
* chronic analgesic use
* diabetes mellitus
* body mass index of (BMI) > 35 kg/m2.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Morphine consumption | postoperative 24 hours
  amount of postoperative 24 hours morphine consumption

SECONDARY OUTCOMES:
Static and dynamic pain score assessed with Numeric Rating Scale (NRS). | postoperative 24 hours
  Pain scores will be noted postoperative at 0, 30 minutes and 1,4,6,12,24 hours. NRS=0 (minimum value, no pain). NRS=10 (maximum value, worst pain imaginable).
intraoperative heart rate | during surgery
  starting from induction to extubation (beat/min)
intraoperative mean arterial pressure | during surgery
  starting from induction to extubation (mmHg)
nause and vomit | postoperative 24 hours
  Assessed with Postoperative Nause and Vomit (PONV) Scale. (0=no PONV, 1=mild nausea, 2=severe nausea or vomiting once, and 3=vomiting more than once)
number of blocked dermatome | 30 minutes after block
  pinprick test in mid-axillar and mid-clavicular line

CONTACTS AND LOCATIONS:
Overall Officials: Nükhet Sivrikoz, Principal Investigator — Attending anesthesiologist
Locations (1):
- Istanbul University, Istanbul Faculty of Medicine, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016